CLINICAL TRIAL: NCT05742646
Title: Managing AsThma AnD Obesity Related Symptoms (MATADORS) Feasibility Study: An mHealth Intervention to Facilitate Symptom Self-management Among Youth
Brief Title: Managing AsThma AnD Obesity Related Symptoms (MATADORS) Feasibility Study
Acronym: MATADORS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00109618; 5P20NR016575-04 (NIH)
Record Dates: First submitted 2023-01-11; First posted 2023-02-24 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Asthma in Children; Obesity; Obesity, Adolescent; Obesity, Childhood
MeSH Terms: conditions — Obesity; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MATADORS app basic information (Active Comparator): The basic app includes real-time symptom monitoring through ecological momentary assessment (EMA) and medication adherence. Basic SMS text messages are sent to participants with reminders to complete EMA questions and enter medication taken. Participants also are provided with activity trackers to assess physical activity and sleep patterns.
  Interventions: Behavioral: MATADORS Control
- MATADORS app to include basic information and expanded educational features (Experimental): Participants in the experimental arm have access to the basic app, along with educational and resource-specific information on asthma, obesity, medications, symptom management, and lifestyle modifications. Features include images, text, and video content. Participants in the experimental arm also are provided with activity trackers to assess physical activity and sleep patterns.
  Interventions: Behavioral: MATADORS

INTERVENTIONS:
Behavioral: MATADORS — Youth will have access to the MATADORS app to include basic information and expanded educational features. They will be asked to log into the app daily for one month and they will be asked to report within the app how they are feeling each day and their medications taken.
  Arms: MATADORS app to include basic information and expanded educational features
Behavioral: MATADORS Control — Youth will have access to the MATADORS app basic information. They will be asked to log into the app daily for one month and they will be asked to report within the app their medications taken.
  Arms: MATADORS app basic information

SUMMARY:
The purpose of this 4 week pilot study is to test the use of a mobile application (also commonly referred to as an app) designed to help increase self-management strategies among youth that have asthma and obesity. The data obtained from this study will facilitate refinement of the app and interventional approaches for a future larger scale study to increase youth self-management of their clinical conditions, symptom management, and health maintenance as they transition to adulthood.

DETAILED DESCRIPTION:
Investigate the feasibility of a 4-week evidence-based, nurse-guided, mHealth self-management intervention application for youth with asthma and obesity (ages 10-17).

Aims are to conduct feasibility testing of the app with a sample of youth randomized to the intervention or control and to obtain estimates of variability and describe preliminary outcomes of the application on fatigue, pain, self-efficacy, anxiety, sleep, depression, and quality of life measured at baseline, 4, and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Youth-Caregiver Dyad Inclusion Criteria:

  * Male and female youth aged 10 - 17 years
  * Adult primary caregiver (18 years and older)
  * English speaking
  * Youth diagnosis of asthma
  * Prescribed inhaler treatment for asthma
  * Youth Body Mass Index at or above the 85th percentile for age and sex based on the Centers for Disease Control (CDC) growth charts
  * Must own a smartphone (iOS) with working Wi-Fi access and/or cellular data plan
  * Prescribed inhaler treatment for asthma

Exclusion Criteria:

* Diagnosis of cognitive impairment
* Inability or unwillingness of youth participant to assent and/or primary caregiver/legal guardian/representative to give informed consent
* Inability or unwillingness to participate in the audio recording interview session or complete study procedures

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Nichols, PhD, RN, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants randomized to control or experimental arms were youth only. Parents reported symptom at baseline and weeks 4 and 8 but were not exposed or involved in other study procedures. Only enrolled youth participated in EMA reports, activity tracking, medication reporting, and engaged with the app. Enrollment numbers represent dyads, although parents weren't not exposed to the intervention regardless of randomization.
Period: Overall Study
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Started | 12 | 12
Youth | 12 | 12
Caregiver | 0 | 0
Completed | 10 | 11
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Baseline data were not collected for caregivers/parents.
Groups:
- MATADORS App Basic Information: MATADORS Control: Youth will have access to the MATADORS app basic information. They will be asked to log into the app daily for one month and they will be asked to report within the app their medications taken. Only youth, not parents, were randomized to control or experimental arms.
- MATADORS App to Include Basic Information and Expanded Educational Features: MATADORS: Youth will have access to the MATADORS app to include basic information and expanded educational features. They will be asked to log into the app daily for one month and they will be asked to report within the app how they are feeling each day and their medications taken. Only youth, not parents, were randomized to control or experimental arms.
- Total: Total of all reporting groups
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 7 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Completing 4-week Study Period
Description: Participant retention and feasibility in completing the 4-week study
Time Frame: 4-week study period
Population: The number of participants analyzed is less than the number enrolled due to loss of follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 10 | 11
Participants | 10 | 11

2. Secondary Outcome: Loss to Follow-up
Description: Number of participants lost to follow-up
Time Frame: 8 weeks
Population: The number of participants analyzed is less than the number enrolled due to loss of follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

3. Secondary Outcome: Study Withdrawals
Description: Number of participants who self withdrew from the study
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 12 | 12
Participants | 2 | 1

4. Secondary Outcome: End of Study Dyadic Interviews
Description: Number of completed end of study dyadic interviews
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 12 | 12
Participants | 7 | 11

5. Secondary Outcome: Change in Fatigue
Description: Change in Fatigue (measured by PROMIS Pediatric Fatigue)-Self-report of fatigue symptoms ranging from tiredness to overwhelming exhaustion. Low score indicates a low level of fatigue and a high score may represent extreme or debilitating levels of exhaustion. Scores above 65 suggest severe fatigue, 55-64 suggest moderate fatigue, 50-54 suggest mild fatigue, and scores less than 50 suggest fatigue scores that are within normal limits (with the lower the number representing healthier rates). 50 indicates the population mean with a standard deviation of 10
Time Frame: 8 weeks
Population: Not all participants completed all end of study surveys.
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 11 | 12
T score
  Baseline | 49 (14.7) | 47.2 (13.8)
  Week 8: number analyzed (Participants) | 10 | 10
  Week 8 | 42.9 (14.1) | 47.2 (12.0)

6. Secondary Outcome: Change in Self-Efficacy
Description: Change in Self-Efficacy (measured by Change in Self-Efficacy for Managing Chronic Disease-6 item scale). This is a 6-item instrument reported on an analog scale that highlights one's confidence in managing their chronic disease. Each item ranges from 1 (minimum; not confident at all) to 10 (maximum; extremely confident). Overall total scores range from 6-60. Minimum total score = 6 and maximum total score = 60. The higher the total score indicates the higher or better level of self-efficacy.
Time Frame: 8 weeks
Population: Not all participants completed all survey instruments at each study visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 11 | 12
units on a scale
  Baseline | 7.4 (1.9) | 7.3 (2.3)
  Week 8: number analyzed (Participants) | 11 | 10
  Week 8 | 8 (1.9) | 7.7 (2.2)

7. Secondary Outcome: Change in Asthma Control
Description: Change in asthma control (measured by Asthma Control Test). Scores range from 5 (poor control of asthma) to 25 (complete control of asthma), with higher scores reflecting greater asthma control. An ACT score >19 indicates well-controlled asthma.
Time Frame: 8 weeks
Population: Instrument administered and analyzed based on chronological age and not all study participants completed surveys at study visits. With MATADORS basic, 11 participants completed baseline and only 10 completed WK8; for the app with expanded features only 11 participants completed baseline and only 10 completed WK 8. a single participant assessed at week 8 was not assessed at baseline, resulting in 12 unique participants analyzed overall
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline 11-12 years old: number analyzed (Participants) | 6 | 6
  Baseline 11-12 years old | 20.8 (4.4) | 20.2 (5.3)
  Baseline 13-17 years old: number analyzed (Participants) | 5 | 5
  Baseline 13-17 years old | 19.2 (5.1) | 16.2 (4.6)
  Week 8 11-12 years old: number analyzed (Participants) | 5 | 6
  Week 8 11-12 years old | 19.6 (5.4) | 20.8 (2.8)
  Week 8 13-17 years old: number analyzed (Participants) | 5 | 4
  Week 8 13-17 years old | 20.6 (2.3) | 17.0 (0)

8. Secondary Outcome: Physical Activity Patterns
Description: Number of minutes active per day
Time Frame: Weekly for 6 weeks (weeks 1-6)
Population: Activity level based on Fitbit data weeks 1-4
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 11 | 12
minutes per day
  Week 1 Very Active | 10.8 (14.6) | 10.4 (11.2)
  Week 2 Very Active | 12.7 (22.0) | 9.3 (10.0)
  Week 3 Very Active | 9.5 (15.1) | 14.6 (15.1)
  Week 4 Very Active: number analyzed (Participants) | 10 | 11
  Week 4 Very Active | 14.1 (19.9) | 14.0 (14.9)

9. Secondary Outcome: Medication Adherence
Description: Self-report of rescue and/or controller medication usage
Time Frame: Daily for 28 days
Population: Outcome data not collected via app as intended due to technological challenges/
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Symptom Reporting
Description: Number of days reporting symptoms of fatigue, pain, anxiety, depression
Time Frame: Daily for 28 days
Population: One control participant did not enter any daily symptom reports.
Measure: Number; unit: Days (cumulative number of days)
Groups:
- MATADORS App Basic Information: MATADORS Control: Youth will have access to the MATADORS app basic information. They will be asked to log into the app daily for one month and they will be asked to report within the app their medications taken and how they are feeling. Only youth, not parents, were randomized to control or experimental arms.
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 11 | 12
Days (cumulative number of days) | 158 | 183

11. Secondary Outcome: Missed School/Work/Activity
Description: Self-report of the number of days where the participant missed school, work, or activities
Time Frame: Baseline, week 4, and week 8
Population: Data not collected via app due to technological uses
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Activity Tracker-step Count
Description: Number of steps taken per day based reported through activity tracker
Time Frame: Daily for 28 days
Population: Daily steps
Measure: Mean (Standard Deviation); unit: Steps per Day
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 11 | 12
Steps per Day
  Week 1 | 3943 (2705) | 5456 (3343)
  Week 2 | 4258 (2941) | 5503 (3317)
  Week 3 | 3683 (3117) | 7294 (3287)
  Week 4: number analyzed (Participants) | 10 | 11
  Week 4 | 5025 (2884) | 6754 (3548)

13. Secondary Outcome: Sleep Patterns
Description: Number of minutes of sleep per day as reported through activity tracker
Time Frame: Weekly for 4 weeks
Population: Daily minutes of sleep times four weeks
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 10 | 12
minutes per day
  Week 1 | 410 (103) | 412 (124)
  Week 2: number analyzed (Participants) | 7 | 8
  Week 2 | 417 (95) | 470 (81)
  Week 3: number analyzed (Participants) | 9 | 10
  Week 3 | 329 (151) | 436 (59)
  Week 4: number analyzed (Participants) | 9 | 9
  Week 4 | 346 (145) | 483 (74)

14. Secondary Outcome: Inability to Concentrate
Description: Self-report on inability to concentrate
Time Frame: Daily for 28 days
Population: Data not collected via app due to technological issues.
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Asthma Belief Survey
Description: The instrument is a 15-item tool that uses a 5-point self-report scale to measure asthma self-efficacy in relation to daily asthma maintenance and an asthma crisis. A rating of 1 = little confidence whereas a rating of 5 = a high confidence level. Responses are averaged across items to indicate an overall score ranging between 1 (low confidence) to 5 (high confidence)
Time Frame: Baseline, week 4, and week 8
Population: Average score 1 (low confidence) to 5 (high confidence)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 11 | 12
score on a scale
  Baseline | 4 (0.7) | 4.1 (0.6)
  Week 4: number analyzed (Participants) | 9 | 11
  Week 4 | 4 (1) | 3.6 (0.9)
  Week 8: number analyzed (Participants) | 10 | 10
  Week 8 | 3.9 (0.8) | 4.2 (0.7)

16. Secondary Outcome: Short Assessment of Health Literacy-English
Description: 18-item instrument to assess the ability to read and understand common medical terms. The total score range is 0-18. A score between 0 and 14 suggests the examinee has low health literacy.
Time Frame: Baseline
Population: Overall score-A score between 0 and 14 suggests the examinee has low health literacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
Number analyzed (Participants) | 12 | 12
score on a scale | 14.2 (2.7) | 14.8 (1.9)

ADVERSE EVENTS:
Time Frame: 4 months
Description: Caregivers were not monitored or assessed for adverse events.
Arm/Group | MATADORS App Basic Information | MATADORS App to Include Basic Information and Expanded Educational Features
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/46/NCT05742646/Prot_SAP_001.pdf
  • Informed Consent Form (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT05742646/ICF_002.pdf